CLINICAL TRIAL: NCT02040025
Title: Evaluating the Effects of EECP on Circulation, Blood Glucose Level and Blood Pressure in Type 2 Diabetes Mellitus
Status: Terminated | Type: Observational
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FDG20140010H
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus
Keywords: hypertension; diabetes mellitus; hemoglobin A1C; peripheral vascular resistance; EECP; Blood pressure; angiogenesis; Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Coronary Artery Disease; Coronary Disease; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this proposed Department of Defense study is to evaluate the effect of Enhanced External Counterpulsation (EECP) on circulation, blood glucose control and blood pressure of type 2 diabetic patients receiving EECP therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or greater than 18
2. Diagnosis of Type 1 or Type 2 diabetes mellitus
3. Prescribed EECP therapy in the DGMC EECP clinic
4. Medically cleared for EECP therapy
5. TRICARE beneficiary

Exclusion Criteria:

1. DGMC EECP clinic patient withou a diagnosis of Type 1 or Type 2 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Defense type 2 diabetic patients enrolled in the Travis AFB, CA EECP clinic.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in TCOM (Transcutaneous oximetry measurement) values | At baseline & post intervention, expected to be on average 30 minutes

SECONDARY OUTCOMES:
Change from baseline in hemoglobin A1C laboratory values | At baseline & post intervention, expected to be on average 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Williams, MD, Principal Investigator — David Grant U.S. Air Force Medical Center
Locations (1):
- David Grant USAF Medical Center, Travis Air Force Base, California, United States

REFERENCES:
- [Background] Martin JS, Beck DT, Aranda JM Jr, Braith RW. Enhanced external counterpulsation improves peripheral artery function and glucose tolerance in subjects with abnormal glucose tolerance. J Appl Physiol (1985). 2012 Mar;112(5):868-76. doi: 10.1152/japplphysiol.01336.2011. Epub 2011 Dec 22. PMID 22194326
- [Background] Bondesson SM, Edvinsson ML, Pettersson T, Edvinsson L. Reduced peripheral vascular reactivity in refractory angina pectoris: Effect of enhanced external counterpulsation. J Geriatr Cardiol. 2011 Dec;8(4):215-23. doi: 10.3724/SP.J.1263.2011.00215. PMID 22783308
- [Background] Braith RW, Conti CR, Nichols WW, Choi CY, Khuddus MA, Beck DT, Casey DP. Enhanced external counterpulsation improves peripheral artery flow-mediated dilation in patients with chronic angina: a randomized sham-controlled study. Circulation. 2010 Oct 19;122(16):1612-20. doi: 10.1161/CIRCULATIONAHA.109.923482. Epub 2010 Oct 4. PMID 20921442